CLINICAL TRIAL: NCT01004406
Title: Plaque Regression and Progenitor Cell Mobilization With Intensive Lipid Elimination Regimen (PREMIER)
Brief Title: Plaque Regression and Progenitor Cell Mobilization With Intensive Lipid Elimination Regimen (PREMIER), Phase I
Acronym: PREMIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLIN-010-09S
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndrome
Keywords: plaque; LDL; statin; endothelial; apheresis; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Plaque, Amyloid | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- intensive LDL-lowering therapy (ILLT) (Experimental): Patient of acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is randomized to LDL-apheresis and an oral daily dose of 40-80mg of Atorvastatin or equivalent
  Interventions: Device: intensive LDL-lowering therapy; Drug: standard statin monotherapy
- standard statin monotherapy (SMT) (Active Comparator): Patient of acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is randomized to an oral daily dose of 40-80mg of Atorvastatin or equivalent without LDL-apheresis
  Interventions: Drug: standard statin monotherapy

INTERVENTIONS:
Device: intensive LDL-lowering therapy — The intensive LDL-lowering therapy uses LDL-apheresis in addition to the standard statin therapy. The device used in this study is the LIPOSORBER LA-15 System, manufactured by Kaneka Pharma America LLC. A filter separates plasma from whole blood, the Liposorber -columns remove LDL from the plasma. The system recombines plasma and blood cells and returns them into the patient's body. This procedure typically takes about 3 hours. The procedure provides an immediate reduction in a patient's lipid levels. A single apheresis treatment can lower LDL by more than 80%, but levels return to baseline within 3 weeks
  Other Names: LIPOSORBER LA-15 System
  Arms: intensive LDL-lowering therapy (ILLT)
Drug: standard statin monotherapy — The standard statin therapy of 40-80mg oral daily dose of Atorvastatin or other equivalent types of statin to lower LDL in blood for both randomized groups.
  Other Names: Atorvastatin or other equivalent types of statin

SUMMARY:
The purpose of this randomized, multi-site, clinical trial is to determine whether intensive therapy consisting of cholesterol-lowering statin drugs plus apheresis to cleanse the blood of low-density lipoprotein (LDL) cholesterol is more effective than statin therapy alone in reducing plaque volume in heart arteries of patients who have already suffered an acute coronary syndrome (ACS). The study will also investigate whether this intensive approach can help increase the presence of endothelial progenitor cells (EPC), stem cells that have been shown to reduce cardiovascular (CV) events in ACS patients. This study has II phases and FDA approval for phase II has been received.

DETAILED DESCRIPTION:
Using statins to lower blood cholesterol, and specifically LDL, is well established as a long-term strategy to reduce CVs and even death. But the most intensive pharmacologic lipid-lowering therapy with statins, though proven superior to standard dose regimens, is still associated with an unacceptably high rate of recurrent CV events early after an ACS. This study hypothesizes that for ACS patients undergoing percutaneous coronary intervention (PCI), intensive lipid-lowering therapy consisting of statins and LDL-apheresis (ILLT) will significantly reduce the total coronary atheroma volume of vulnerable plaque and augment mobilization of peripherally circulating EPC colony forming units, compared to guideline statin monotherapy (SMT). ILLT will lead to fewer CV events for these patients.

Patients presenting at two VA sites with ACS will be screened and consented before undergoing uncomplicated PCI (balloons or stents) and intravascular ultrasound with virtual histology (IVUS-VH). They will then be randomized into the ILLT arm or SMT arm of the study. The ILLT group will receive one treatment of LDL-apheresis plus a daily oral 80mg dose of Atorvastatin; the SMT group will only get the Atorvastatin. Patients will again undergo IVUS-VH 12 weeks after enrollment to measure atheroma volume; EPC level will also be checked.

The four-year duration of the study includes 24 months of accrual, six months of follow-up, and 12 months of study closure and data analysis. A two-sample t-test of mean difference with 90% power and 0.65 Cohen's D effect size provides a total sample size estimate of 102. Counting 20% drop-out rate, the sample size increases to 128.

The recent FDA recommendations regarding the design of the study has been included in the revised study protocol:

1. The first stage will enroll 30 patients with a 2:1 randomization favoring LDL-apheresis. the safety data will be submitted to the FDA.
2. The enrollment of the second stage of the study will be contingent to the recommendations of the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent (including HIPAA)
* Age >30 years
* Presenting with acute coronary syndrome (ACS), manifested as unstable angina or non-ST-elevation myocardial infarction
* Referred for clinically-indicated, non-emergent (the procedure is not required to be performed within 3 hours after patient presentation) coronary angiography and PCI with IVUS-VH of target coronary artery for ACS
* Successful placement of two large bore IV cannulas in bilateral upper extremities
* Fasting (>= 12 hours) LDL >= 100mg/dl while on <= 80mg Atorvastatin or equivalent dose of other statin, performed at time of admission or 3 months prior to PCI.

Exclusion Criteria:

* Known allergy to aspirin, clopidogrel, statins, or iodinated contrast
* Positive pregnancy test, planning to become pregnant, or breast-feeding
* Coexisting conditions that limit life expectancy to less than six months or affect patient compliance
* Uncontrolled fasting (>= 12 hours) triglyceride levels (>= 500mg/dl)
* Already participating in an investigational device or drug study
* History of heparin induced thrombocytopenia (HIT)
* Persons with estimated glomerular filtration rate (eGFR) less than 60 ml/min if they are diabetic; persons with eGFR of less than 45 ml/min if they are not diabetic
* ST-elevation myocardial infarction at admission
* Abnormal liver function test (LFT) at time of admission or 3 month prior to PCI with abnormal LFT defined as any liver transaminases (ALT or AST) 3 times the upper limit of the normal laboratory reference
* Pre-PCI or post-PCI left ventricular ejection fraction <25% by echo or cardiac catheterization done after admission
* Pre-PCI, intra-PCI, or post-PCI hemodynamic instability with hypotension
* Pre-PCI, intra-PCI, or post-PCI cardiac arrest
* Pre-PCI or post-PCI heart failure with or without pulmonary edema
* Intra-PCI or post-PCI sustained ventricular tachycardia
* Complicated PCI, defined as PCI with any of the vascular access complications (large hematoma with lump > 5 cm or requiring medical treatment; arteriovenous (AV) fistula; pseudo aneurysm requiring treatment; retroperitoneal bleeding), or PCI with any of the procedural complications (abrupt vessel closure; no-reflow phenomenon; new angiographic thrombus; new major dissection with reduced flow; catheter-related thrombus), or PCI requiring further medical treatments (urgent coronary artery bypass grafting (CABG); endotracheal intubation; unplanned in-aortic balloon pump; left ventricular assist device (LVAD); covered stent; unplanned temporary pacemaker wire; administration of inotropes; CPR) , or PCI resulting in clinical events (death; stroke; myocardial infarction; stent thrombosis) during or within 24 hours after the index PCI
* Post-PCI ongoing chest pain
* Post-PCI severe groin pain and hematoma > 5cm in diameter
* Persons whose hemoglobin is less than 9 grams following the index PCI/IVUS procedure, or who experience a drop in hemoglobin of greater than or equal to 2 grams following the procedure
* Not able to comply with study protocol as determined by the investigators

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — VA North Texas Health Care System, Dallas
Locations (2):
- United States (2):
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA North Texas Health Care System, Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee S, Luo P, Reda DJ, Latif F, Hastings JL, Armstrong EJ, Bagai J, Abu-Fadel M, Baskar A, Kamath P, Lippe D, Wei Y, Scrymgeour A, Gleason TC, Brilakis ES. Plaque Regression and Endothelial Progenitor Cell Mobilization With Intensive Lipid Elimination Regimen (PREMIER). Circ Cardiovasc Interv. 2020 Aug;13(8):e008933. doi: 10.1161/CIRCINTERVENTIONS.119.008933. Epub 2020 Aug 14. PMID 32791950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment for Phase I pilot study started on September 6, 2011, and the first participant was randomized on September 8, 2011. The recruitment period stopped in June 2012. For 2 participating sites, Dallas and Oklahoma City randomized 26 and 5 participants, respectively.
Pre-assignment Details: There were 59 subjects consented and enrolled into the study before entering catheterization lab to have the PCI procedure, but 28 subjects were not randomized to treatment assignments with the major exclusion reasons as not referred for PCI or not able to comply with study protocol based on the inclusion/exclusion criteria.
Groups:
- Intensive LDL-lowering Therapy (ILLT): Patient of acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is randomized to LDL-apheresis in addition to the standard statin therapy of an oral daily dose of 40-80mg of Atorvastatin or equivalent. The device used in this study is the LIPOSORBER LA-15 System, manufactured by Kaneka Pharma America LLC. A filter separates plasma from whole blood, the Liposorber -columns remove LDL from the plasma. The system recombines plasma and blood cells and returns them into the patient's body. This procedure typically takes about 3 hours. The procedure provides an immediate reduction in a patient's lipid levels. A single apheresis treatment can lower LDL by more than 80%, but levels return to baseline within 3 weeks.
Period: Overall Study
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Started | 21 | 10
Completed | 18 | 10
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT) | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (6.9) | 57.6 (7.7) | 61.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 10 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 7 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 10 | 31
Weight [Mean (Standard Deviation); unit: pounds] | 207.8 (28.9) | 211.4 (38.8) | 208.9 (31.8)
Height [Mean (Standard Deviation); unit: inches] | 69.5 (2.7) | 71.0 (2.0) | 70.0 (2.6)
Heart Rate [Mean (Standard Deviation); unit: beats/min] | 76.9 (11.2) | 76.3 (7.2) | 76.7 (10.0)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 144.0 (26.2) | 150.1 (23.6) | 145.9 (25.2)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 80.8 (14.0) | 85.3 (14.4) | 82.3 (14.1)
Smoker [Count of Participants; unit: Participants]
  Never | 6 | 4 | 10
  Current | 6 | 3 | 9
  Former | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total Atheroma Volume of the Target Coronary Artery From Baseline to 12 Weeks Post-PCI as Assessed Via Intravascular Ultrasound With Virtual Histology (IVUS-VH)
Description: The primary effectiveness outcome measure was the change in the total atheroma volume within a ≥ 20 mm long segment of the target coronary artery from baseline to 12 weeks post-PCI. The measurement was done via IVUS-VH at 2 time points (baseline during index PCI and 12-week follow-up).
Time Frame: baseline and 12-week follow-up
Population: Reported results are based on Intent-to-Treat (ITT) approach.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 21 | 10
mm^3 | -3.70 (18.52) | 10.79 (35.23)

2. Secondary Outcome: Change in % Necrotic Core (NC) Component of Atheroma From Baseline to 12 Weeks Post-PCI as Assessed Via IVUS-VH
Description: The %NC component of atheroma were obtained via IVUS-VH at 2 time points (baseline during index PCI and 12-week follow-up).
Time Frame: baseline and 12-week follow-up
Population: Reported results are based on ITT approach.
Measure: Mean (Standard Deviation); unit: percentage of atheroma component
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 21 | 10
percentage of atheroma component | 0.007 (0.03) | -0.006 (0.03)

3. Secondary Outcome: Endothelial Progenitor Cell Colony Forming Units (EPC-CFU) Per Milliliter of Peripheral Blood Across Time
Description: The cell culture assay and quantification of circulating EPC-CFU were performed for patients recruited at the Dallas VA center only. The assay were done at 4 time points (pre-PCI, post-PCI, 4-week follow-up, and 12-week follow-up).
Time Frame: pre-PCI, post-PCI, 4-week follow-up, and 12-week follow-up
Population: Reported results are based on observed data from participants who had secondary outcome measured. This outcome was captured for Dallas site only.
Measure: Mean (Standard Deviation); unit: colonies/ml
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 16 | 9
colonies/ml
  baseline pre-PCI | 13.71 (6.53) | 13.89 (4.94)
  baseline post-PCI | 15.85 (6.40) | 13.33 (4.29)
  4-week follow-up | 25.39 (10.31) | 17.86 (8.91)
  12-week follow-up | 27.62 (12.59) | 21.50 (9.84)

4. Secondary Outcome: Major Adverse Cardiovascular Events
Description: The number of patients who experienced major adverse cardiovascular endpoints (MACE) including death, myocardial infarction, coronary revascularization, and stroke during the follow-up periods.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 21 | 10
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AE), Serious Adverse Events (SAE), and Unanticipated Adverse Device Effects (UADE) were monitored at the study sites throughout the whole period of the study at each clinic visit and telephone contact, beginning as soon as a study participant signs the Informed Consent and continuing through end-of-study for each participant. Most participants were followed for around 6 months for AE/SAE/UADE.
Description: All AE/SAE/UADE including both those related to the study intervention and those not related to the intervention, will be collected and recorded on the appropriate case report forms (CRF). For the purpose of safety monitoring, the study intervention is defined as the use of 1) statins with or without the addition of LDL-apheresis, 2) LDL-apheresis, and 3) cardiac catheterization and IVUS-VH as described in this protocol.
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 10/21 | 4/10
Other Adverse Events (participants affected / at risk) | 17/21 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive LDL-lowering Therapy (ILLT) (N=21) | Standard Statin Monotherapy (SMT) (N=10)
Chest pain (General disorders) | 3 (3) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive LDL-lowering Therapy (ILLT) (N=21) | Standard Statin Monotherapy (SMT) (N=10)
Chest pain (General disorders) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Our study is limited by its relatively small sample size and short follow-up. All study sites were Veterans Affairs medical centers and therefore enrolled a disproportionate number of men, limiting the generalizability of its findings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes